CLINICAL TRIAL: NCT06490016
Title: Effect of Web Based Menstrual Health Education on Menstrual Attitude, Menstrual Symptoms and Anxiety Among Visually Impaired Adolescent
Brief Title: Menstrual Health Education for Visually Impaired Adolescent
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, hatice güdül öz, Research Assistant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 04.02.2023/83; 223K208 (Other Grant/Funding Number: TUBITAK 1001)
Record Dates: First submitted 2024-06-14; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Visual Impairment; Menstrual Problem
Keywords: anxiety; health education; nurse; menstruation; visually impaired adolescent
MeSH Terms: conditions — Vision Disorders; Menstruation Disturbances; Anxiety Disorders; Health Education

STUDY DESIGN:
Intervention Model Description: There are 2 groups: 2 interventional group
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group that given face to face education (Experimental): 6 face-to-face meetings will be held with adolescent disabled girls. Training will be held collectively at school or in an association. The training modules will last 3 weeks and 5 modules will be used in the training. (1st Meeting and Survey collection, 2nd week: 1st and 2nd module, 3rd week: 3 modules and 4th week: 5 modules, 6th interview: after training). Training modules will be given every week at a determined place and time. Following the training, the effect of the training will be investigated by repeating the data collection forms twice at 1-month intervals during the menstrual periods of the participants.
  Interventions: Behavioral: Face to face
- Intervention group that given web-based education (Experimental): This group will not be met face to face and communication will be provided via the website. A username and password will be defined for each user before entering the web page. Visually impaired adolescent girls will be able to individually enter the relevant modules without assistance, read the module they want, and listen to the depicted pictures and graphics. From the admin section of the website, it will be tracked who attended the training, how many minutes they stayed, and how many times a week they attended. The training modules will last 3 weeks and 5 modules will be used in the training. (1st Meeting and Survey collection, 2nd week: 1st and 2nd module, 3rd week: 3 modules and 4th week: 5 modules, 6th interview: after training). A reminder notification will be sent to the contact section on the website every week for them to attend the training.
  Interventions: Device: web based education

INTERVENTIONS:
Device: web based education — The web page will be prepared with professional support in line with the guidelines of the Web Content Accessibility Guide (WCAG / WIEK 2.1) developed by W3C.
  1. st meeting: online "Informed Consent" will be obtained. After the meeting, the Personal Information Form, Menstrual Attitude Scale, Menstrual Symptom Scale, State and Trait Anxiety Scale will be filled out online.
  2. nd interview: Module 1-2.
  3. rd interview: Module 3 -4.
  4. th meeting: Module 5.They will be asked to fill out the System Usability Scale.
  5. th interview: During the first menstrual period after the training, the Menstrual Attitude Scale, Menstrual Symptom Scale, and State Anxiety Scale will be completed online.
  6. th interview: During the second menstrual period after the training, the Menstrual Attitude Scale, Menstrual Symptom Scale, and State Anxiety Scale will be completed online.
  Arms: Intervention group that given web-based education
Behavioral: Face to face — In face-to-face training, "female internal reproductive organ models", "female external reproductive organ models", "training content prepared with Braille alphabet", "menstrual hygiene management kit (underwear, pads, napkins, calendar)" materials will be used. Pictures and audio descriptions will be used in web-based training.
  1. st interview: "Informed Consent" . After the meeting, the Personal Information Form, Menstrual Attitude Scale, Menstrual Symptom Scale, State and Trait Anxiety Scale will be filled out.
  2. nd meeting: Module 1-2
  3. rd meeting: Module 3- 4
  4. th meeting: Module 5.
  5. th interview: Menstrual Attitude Scale, Menstrual Symptom Scale, State Anxiety Scale will be completed.
  6. th interview: Menstrual Attitude Scale, Menstrual Symptom Scale, State Anxiety Scale will be completed.
  Arms: Intervention group that given face to face education

SUMMARY:
This study was planned as a two-group randomized controlled interventional study to determine the effect of face-to-face and web-based menstrual health education given to visually impaired adolescent girls on menstrual attitude, menstrual symptoms and anxiety.

DETAILED DESCRIPTION:
Menstruation is a physiological and natural process of the reproductive system. It is reported that more than 300 million individuals menstruate every day worldwide. On average, a woman menstruates for approximately 3,000 days, or 8 years, between the ages of 11 and 49. Therefore, menstruation is an important issue that requires physical, spiritual and social adaptation for women. It is known that the majority of menstruating individuals have serious problems in managing their monthly menstrual cycles healthily and effectively. However, the menstrual needs of girls and women with different types of disabilities vary compared to individuals without disabilities.

Since the sense of sight has an important place in performing daily activities, visually impaired girls and women are one of the disabled groups that experience various difficulties during the menstrual process. In the literature, it is seen that visually impaired individuals have negative myths and beliefs about the menstrual period, have difficulties with self-care, do not comply with hygiene rules during the menstrual period, and talk about menstrual hygiene management with their mothers, sisters, friends, etc. It is emphasized that there are deficiencies in their knowledge and practices regarding menstrual hygiene, that they see the menstrual period as a shame, and that they experience difficulties such as social isolation and forced sterilization. In this context, the menstrual period emerges as an important global public health problem for visually impaired girls and women.

Menstrual health/hygiene management is important in order to cope with the problems experienced during menstruation. United Nations International Children's Emergency Fund underlines that menstrual health and hygiene management should be addressed within a broader framework, reconciling health, well-being, gender equality, education, social equality, individual empowerment policies and human rights. The only point that distinguishes visually impaired women from sighted women regarding menstruation is menstrual hygiene management. Menstrual management in visually impaired women; It varies depending on the use of materials such as pads and tampons, hygiene training, degree of social support, disability status of the person and symptoms related to menstruation. Different methods and tools can be used in training for visually impaired individuals. When providing education to visually impaired individuals, changes should be made in the tools used rather than the content of the education. Because lack of vision does not constitute an obstacle to their education. Training can be provided using models, printed brochures containing the Braille alphabet, voice recordings and assistive technologies.

The comprehensive menstrual hygiene management training to be prepared will guide health professionals, special education teachers and institutions. Studies have reported that nurses have difficulty and experience communication problems while providing care to disabled individuals. It is believed that it will guide nurses regarding the educational methods and needs of visually impaired individuals. In addition, it is a study that can support healthcare personnel who may be inadequate in consultancy and training roles due to the insufficient number of healthcare personnel in our country and their high workload. In particular, the widespread use of web-based training in the education of disabled individuals can be an opportunity for many disabled individuals who have economic, transportation and material problems, regardless of time and place.

Hypotheses of the research:

Ho: Between groups; Ho1: There is no difference between menstrual attitude scale scores in web-based and face-to-face menstrual health education.

Ho2: There is no difference between menstrual symptom scale scores in web-based and face-to-face menstrual health education.

Ho3: There is no difference between anxiety scores in web-based and face-to-face menstrual health education.

H1: Between groups:

H11: There is a difference between menstrual attitude scale scores in web-based and face-to-face menstrual health education.

H12: There is a difference between menstrual symptom scale scores in web-based and face-to-face menstrual health education.

H13: There is a difference between anxiety scores in web-based and face-to-face menstrual health education.

ELIGIBILITY:
Inclusion Criteria:

* For face-to-face education:

  * Be between the ages of 11-19
  * Ability to read and write
  * Menstruation
  * Having at least 60% vision loss (those with congenital or acquired vision loss)

For web-based training:

* Be between the ages of 11-19
* Ability to read and write
* Menstruation
* Having at least 60% vision loss (those with congenital or acquired vision loss)
* Having a computer or mobile phone compatible with a screen reader program and internet access.

Exclusion Criteria:

• Not attending face-to-face or web-based training for at least 1 week.

Ages: 11 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure 1 | during 6 week
  Menstrual Attitude Scale will be used to score the menstrual attitude level. The scale consists of 33 items. MBI consists of five subscales that question the positive and negative aspects of menstruation.
  1. Menstruation as a debilitating phenomenon,
  2. Menstruation as a disturbing phenomenon,
  3. Menstruation as a natural phenomenon,
  4. Noticing/anticipating that menstruation will occur
  5. Deny the effects of menstruation. The scale is Likert type and evaluated between 1-7. The reliability coefficient of the original scale is 0.95-0.97. A high average of the scores obtained from the items, subgroups or the entire scale in the Menstruation Attitude Scale indicates that the attitude towards menstruation is "positive". As the scores of the scale increase, the positive attitude towards menstruation increases.
  At the same time, it is planned to increase the scale score by providing planned training.
Primary Outcome Measure 2 | during 6 week
  The Menstrual Symptom Scale will be used to score menstrual symptom level.
  The Menstruation Symptom Scale evaluates menstrual pain and symptoms. Participants are asked to give a number between 1 (never) and 5 (always) to the symptoms they experience regarding menstruation. 1-13. Items belong to the "Negative effects/somatic complaints" subscale, items 14-19. The items refer to the "Menstrual pain symptoms" subscale and items 20-22. The items belong to the "Coping methods" sub-dimension. Cronbach's Alpha value is 0.86. It is a five-point Likert type scale consisting of 22 items. The score obtained from the sub-dimensions is calculated by taking the total score average of the items in the sub-dimensions. An increase in the mean score for sub-dimensions indicates that the severity of menstrual symptoms related to that sub-dimension has increased.
  At the same time, it is planned to reduce the scale score by providing planned training.
Primary Outcome Measure 3 | during 6 week
  State and Trait Anxiety Scale will be used to score the state and trait anxiety level.
  Each expression in the scale is "Not at all" (1), "Somewhat" (2), "A lot" (3), "Completely" (4). It indicates that 0-19 points obtained from the scale mean no anxiety, 20-39 points mean mild anxiety, 40-59 points mean moderate anxiety, and 60-79 points mean severe anxiety, and individuals with scores of 60 and above need professional help.
  At the same time, it is planned to reduce the scale score by providing planned training.

CONTACTS AND LOCATIONS:
Overall Officials: Evşen Nazik, PhD,RN, Study Director — Cukurova University
Locations (1):
- Çukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No